CLINICAL TRIAL: NCT01133184
Title: The Employing of the Bio-Hep-B PreS1/PreS2/S Hepatitis B Virus (HBV) Vaccine in New Born Babies From HBV Positive Palestinian Mothers
Brief Title: Improved Prevention of Perinatal Hepatitis B Transmission
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Rifaat Safadi, Hadassah Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 0509-08-HMO
Record Dates: First submitted 2010-05-25; First posted 2010-05-28 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-01

CONDITIONS: Liver Fibrosis
Keywords: HBV transmission PreS1/PreS2/S HBV vaccine
MeSH Terms: conditions — Liver Cirrhosis | interventions — Pre-S vaccine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Sci B vac — Sci B vac

SUMMARY:
Impaired activity of Natural Killer (NK) cells has been proposed as a mechanism contributing to viral persistence in Hepatitis C Virus (HCV) infection. NK cells display anti-fibrotic activities by killing activated hepatic stellate cells (HSCs) that have lost the self-recognition marker; Major Histocompatibility (MHC) class I. Determining the down-expressed genes on NK cells necessary for their anti-fibrotic activity was never studied previously. This will allow us to study their role fully in phagocytosis process as well as their interaction of HSCs and therefore manipulating these genes using molecular techniques. Exploring the cellular functions of these genes will highlight their involvement in the progression of liver fibrosis and could be used as a therapeutic tool for preventing the disease.

DETAILED DESCRIPTION:
Lymphocyte/Hepatic stellate cells (HSCs) interactions via adhesion and phagocytosis are mediated as well as affected among others by Leptin, Endocannabinoids (CB) receptors, adiponectin, progesterone as well as by number of CD8 and NK related adhesion/phagocytosis candidate genes. Those pathways may explain the impaired activity of NK cells in Hepatitis C Virus (HCV)cirrhotic cases.

In this perspective, we propose the following specific aims:

1. To confirm by repeated gene arrays the pro/anti-fibrotic genes expressed by NK and CD8 lymphocyte-subsets in human healthy volunteers and patients with HCV cirrhosis. Then to explore the same issue of lymphocyte gene array (NK and CD8 cells) in naïve and carbon tetrachloride fibrosis model in mice. Then to support results by the Real Time PCR and conduct bio-informatics assessments of results.
2. Evaluate the role of Leptin, CB receptors and adiponectin in the lymphocyte/HSCs phagocytosis process. This would be tested both by in-vitro and in-vivo settings using cell cultures and knock-out mice (CB2-/-, Adiponectin-/- and leptin-/-Ob/Ob). The use of lymphocyte adoptive transfer model with immune manipulations will guide us for a specific functional role of each target gene in the specific lymphocyte subset.
3. To evaluate how lymphocyte/HSC phagocytosis process affected by other CD8 and NK related gene candidates extrapolated from the results of earlier aims (see preliminary data). Suggested genes are including: Immune synapse genes (CHST13 and NLGN4X) to obtain the expected anti-fibrotic response. Genes with HSCs phagocytotic activity that is providing possible pathways for the HCV related escape from the expected anti-fibrotic response and eventually pro- fibrotic consequences (AIF1, CHST13, hnRPL). Killer cell lectin-like receptor subfamily C, member 2 (NKG2C; CD159c) is down expressed over HCV related CD8 cells suggesting a decrease of HSCs killing by the CD8 cells. Progestin & adipoQ receptor family member IV (PAQR4): Progesterone and adipoQ receptors are down-expressed over HCV related CD8 cells. Adiponectin is anti-fibrogenic mediator and is a candidate as PAQR4 ligand. When PAQR4 receptor is down- regulated in CD8 cells, it is suggested that this would be a mechanism for immune impairment. Also, Moreover, Progesterone and adipoQ receptors down- expression is supporting our mice animal model results that pregnancy caused progression of hepatic fibrogenesis associated with increased CD8 subsets and NK-T cells. We are going to evaluate the specific effect in the phagocytosis process.
4. To evaluate if HCV by itself or HCV related proteins are directly responsible for the NK related impairment. Transgenic mice for the HCV envelop proteins will be used to assess alterations of lymphocyte subsets and phagocytosis ability.

The expected results will extend the knowledge of hepatic fibrogenesis in particular but may provide more application in general immunology. Therefore, expected results will be potentially a new target for anti-fibrotic designs and possibly in other medical conditions. Not only liver cirrhosis will be potentially prevented following anti-fibrotic therapies but also the hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

* All Hepatitis B s Antigen (HBsAg) positive pregnant women attending the centers will be suggested to participate in the study and therefore provided with all information needed

Exclusion Criteria:

* Co-infection with HIV
* Mothers with immune suppression

Max Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6343 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-03 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Co-infection with Hepatitis D and HIV. | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Rifaat Safadi, M.D, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

REFERENCES:
- [Derived] Safadi R, Khoury T, Saed N, Hakim M, Jamalia J, Nijim Y, Farah N, Nuser T, Natur N, Mahamid M, Amer J, Roppert PL, Gerlich WH, Glebe D. Efficacy of Birth Dose Vaccination in Preventing Mother-to-Child Transmission of Hepatitis B: A Randomized Controlled Trial Comparing Engerix-B and Sci-B-Vac. Vaccines (Basel). 2021 Apr 1;9(4):331. doi: 10.3390/vaccines9040331. PMID 33915943